CLINICAL TRIAL: NCT04595591
Title: Effects of Propofol Titration at Different Speeds on Hemodynamics and Stress During General Anesthesia Induction
Brief Title: Observation of Propofol Titration at Different Speeds
Acronym: OPTDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SanQing Jin (Other)
Responsible Party: Sponsor-Investigator, SanQing Jin, professor, Sixth Affiliated Hospital, Sun Yat-sen University
Organization: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020ZSLYEC-182
Record Dates: First submitted 2020-09-23; First posted 2020-10-20 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia, General; Hemodynamics
Keywords: titration of propofol
MeSH Terms: interventions — Remifentanil; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Ⅰ (Active Comparator): titration dosing speeds of propofol at 2mg/kg/min
  Interventions: Drug: 2mg/kg/min
- Group Ⅱ (Active Comparator): titration dosing speeds of propofol at 1mg/kg/min
  Interventions: Drug: 1mg/kg/min
- Group III (Active Comparator): titration dosing speeds of propofol at 0.5mg/kg/min
  Interventions: Drug: 0.5mg/kg/min

INTERVENTIONS:
Drug: 2mg/kg/min — titration dosing speeds of propofol at 2mg/kg/min
  Other Names: Remifentanil 2ug/kg; Rocuronium 1.5mg/kg
  Arms: Group Ⅰ
Drug: 1mg/kg/min — titration dosing speeds of propofol at 1mg/kg/min
  Other Names: Remifentanil 2ug/kg; Rocuronium 1.5mg/kg
  Arms: Group Ⅱ
Drug: 0.5mg/kg/min — titration dosing speeds of propofol at 0.5mg/kg/min
  Other Names: Remifentanil 2ug/kg; Rocuronium 1.5mg/kg
  Arms: Group III

SUMMARY:
Propofol is one of the most widely used anesthetics for its fast onset and quick elimination. The conventional speed of its induction dose often causes severe hemodynamics fluctuations with hypotension and arrhythmia. The recommended dosage on the drug insert comes from group pharmacokinetic studies which does not apply to the specific situation of every patient, so the investigators emphasize individualized medication. The investigators have observed the titration of propofol in general anesthesia induction, and found that the dosage was less and the hemodynamics was becoming more stable. At the same time, the investigators found that the hemodynamics still has obvious fluctuations in the titration of the administration rate recommended in the instructions. The investigators intend to further compare the effects of propofol titration administration at different rates for hemodynamics and stress during the induction period of general anesthesia, and find a safer and more appropriate rate of administration.

DETAILED DESCRIPTION:
Based on the recommended dosing speed in the propofol instructions, this research protocol further reduces the dosing speed (40 mg administered every 10 seconds), and sets three different titration dosing speeds: group I 2 mg/kg/min; group II 1 mg /kg/min; group III 0.5 mg/kg/min. The program is calculated by statistics, and it will be planned to enroll 276 participants undergoing elective surgery under general anesthesia with oral endotracheal intubation, and randomly divided into 3 groups according to a random number table, with 92 cases in each group. When participants reach the titration endpoint (OAAS score 1 point) during the titration of propofol in the induction, the investigators stop the dosing and switch to a maintenance dose, and give rocuronium 0.15 mg/kg and remifentanil 2 ug/kg; 2 minutes later the chief anesthetist performs tracheal intubation. The investigators will observe hemodynamics changes and brain electrical activity throughout the process, and adjust the drugs according to the blood pressure to make the hemodynamics as stable as possible.

After confirming the successful tracheal intubation, the investigators will give participants machine-controlled ventilation, and the total intravenous anesthesia (TIVA) will be given with propofol, remifentanil, and cis-atracurium. During the operation, remifentanil will be injected with a constant rate of 0.2ug/kg/min, and propofol will be injected with a fluctuating rate of 2-8mg/kg/h (the pump injection rate will be adjusted according to blood pressure and BIS, and the rate of remifentanil can be adjusted if necessary) to maintain BIS between 40-60.Fluid therapy will be performed according to the participants' hemodynamics and intraoperative conditions. After extubation, participants will be sent to the postoperative recovery room; a follow-up visit will be performed the next day, and a telephone return visit will be performed on the 30th day.

The investigators record the visual analogue scale(VAS) score for preoperative anxiety of each participant, bispectral index (BIS) and hemodynamics of patients when participants reach different stages of sedation as determined by the Observer's Assessment of Alertness/Sedation Scale (OAAS) score, and the lowest value and specific time of mean blood pressure(MBP) and BIS during induction of anesthesia；the investigators record various parameters at the following time points(10 minutes after entering the operating room before propofol administration, every minute after administration until intubation, immediately after tracheal intubation, and 1, 2, 4, 6, 8, 10, 20 min after intubation), and parameters include: systolic blood pressure(SBP) , diastolic blood pressure(DBP), MBP, heart rate(HR), electrocardiogram ST-T changes (V1), BIS, cardiac function parameters (heart rate variability(HRV), stroke volume (SV), stroke index(SVI), cardiac output (CO), cardiac index(CI) ), oxygen delivery parameters (oxygen delivery (DO2), oxygen delivery index (DO2I)), peripheral vascular resistance parameters (systemic vascular resistance (SVR), systemic vascular resistance index (SVRI)), volume parameters (stroke volume variation(SVV), pulse pressure variation (PPV), increase in stroke volume(△SV)); the investigators record the time for each participant reach the titration endpoint and the amount of propofol used, the time from the start of induction to the completion of the tracheal intubation and the amount of propofol, and the total amount of propofol during the operation.

The investigators record invasive blood during the trial, and use cameras to video the entire process of anesthesia induction.

The 11-30th participants in each group will be given arterial blood samples at 1, 3, 5, and 7 minutes after the administration of propofol to measure the blood concentration of propofol; when rocuronium is given and 30 seconds after the completion of tracheal intubation, venous blood will be drawn to measure the catecholamine concentration; ten cases of propofol with high, medium and low sensitivity will be selected for transcriptome RNA sequencing; Single nucleotide polymorphism（SNP） analysis of propofol-related genes in special cases.

During the induction period, the investigators will monitor EEG of the left and right frontal, temporal and occipital lobes, and analyze the power spectrum of β, α, θ, and σ brain waves; observe the pupil reflex and auditory evoked potential(brain stem auditory evoked potentials(BAEP): the incubation period and amplitude of III, V ; middle latency auditory evoked potentials（MLAEP）: the incubation period and amplitude of Pa, Nb) before induction , when the titration endpoint reaches and after finishing intubation.

Blind design:

The observer performs pre-entry screening, and does not know the group of participants during the induction process. The anesthesia nurse receives the experiment envelope in advance, adjusts the infusion pump according to the group, and adjusts the pump to the position facing away from the observer and the chief anesthetist. The chief anesthetist communicates with patients and performs OAAS scores scoring. When the titration endpoint reaches, the anesthesia nurse will stop propofol administer and shift to the maintenance dose, following the observer's order to add vasoactive drugs or propofol during the induction process, and do not participate in the postoperative follow-up work. The chief anesthetist (working for more than 3 years) is responsible for assisted ventilation and tracheal intubation. The anesthesiologist in the resuscitation room, the patient, and the post-operative return visitor do not know the group of the participant.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 Years old
2. Elective surgery for general anesthesia through oral tracheal intubation and surgery is expected to last more than 2 hours
3. The American Society of Anesthesiologists(ASA) grade is I or II, and the cardiac function is 1-2;
4. Body mass index (BMI) 18-30 kg/m2;

Exclusion Criteria:

1. Patients have severe heart, lung, liver, and kidney diseases (heart function grade>3 / respiratory failure / liver failure / renal failure)
2. Patients with arrhythmia: sinus bradycardia (ventricular rate <60 beats/min), atrial fibrillation, atrial flutter, atrioventricular block, frequent ventricular premature, multi-source ventricular premature, ventricular premature R on T, Ventricular fibrillation and ventricular flutter.
3. Patients who are expected to be difficult to intubate, hypoalbuminemia(albumin is less than 35g/L), hypertension and diabetes;
4. Patients with a higher risk of reflux and aspiration, such as full stomach, gastrointestinal obstruction, gastroparesis, and pregnant women;
5. Patients have schizophrenia, epilepsy, Parkinson's disease, intellectual disability, hearing impairment, abnormal EEG, etc.;
6. Patients who take sedative and analgesic drugs for a long time;
7. Patients who are allergic to propofol or its fat emulsion;
8. Patients who are participating in other clinical trials, and who refuse to sign informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 276 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-25 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure(MBP) | During the procedure of anesthesia induction
  Relative change of MBP(decreased more than 30%) in the three groups

SECONDARY OUTCOMES:
Stroke Volume (SV) | During the procedure of anesthesia induction
  Relative change of SV (ml/beat) in the three groups
Cardiac Output (CO) | During the procedure of anesthesia induction
  Relative change of CO (litre/min) in the three groups
Systemic Vascular Resistance (SVR) | During the procedure of anesthesia induction
  Relative change of SVR (dynes-sec/cm5/m2) in the three groups
Catecholamine | During the procedure of anesthesia induction
  Concentration of catecholamines in venous blood before and after tracheal intubation in the three groups
Plasma concentration change curves | During the procedure of anesthesia induction
  Plasma concentration change curves of propofol in the three groups
The relative level of mRNA in serum | Baseline
  Expression differences of RNA sequences in groups of high, middle and low propofol sensitivity through bioinformatics analysis.
Brain electrical activity | During the procedure of anesthesia induction
  Differences of brain electrical activity (EEG, AEP)in the three groups
The dosage of propofol | Through anesthesia completion, an average of 3 hours.
  The dosage of propofol (reach the end of the titration, complete the tracheal intubation ) and intraoperative maintenance dosage in the three groups
Induction time | Through anesthesia completion, an average of 3 hours.
  Induction time in the three groups
Recovery time | Through anesthesia completion, an average of 3 hours.
  Postoperative recovery time in the three groups
The occurrence of important cardiovascular events | One month after finish operation
  The occurrence of important cardiovascular events during the perioperative period

CONTACTS AND LOCATIONS:
Overall Officials: SanQing Jin, MD, Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- the Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jor O, Maca J, Koutna J, Gemrotova M, Vymazal T, Litschmannova M, Sevcik P, Reimer P, Mikulova V, Trlicova M, Cerny V. Hypotension after induction of general anesthesia: occurrence, risk factors, and therapy. A prospective multicentre observational study. J Anesth. 2018 Oct;32(5):673-680. doi: 10.1007/s00540-018-2532-6. Epub 2018 Jul 19. PMID 30027443
- [Background] de Wit F, van Vliet AL, de Wilde RB, Jansen JR, Vuyk J, Aarts LP, de Jonge E, Veelo DP, Geerts BF. The effect of propofol on haemodynamics: cardiac output, venous return, mean systemic filling pressure, and vascular resistances. Br J Anaesth. 2016 Jun;116(6):784-9. doi: 10.1093/bja/aew126. PMID 27199311
- [Background] Walsh M, Devereaux PJ, Garg AX, Kurz A, Turan A, Rodseth RN, Cywinski J, Thabane L, Sessler DI. Relationship between intraoperative mean arterial pressure and clinical outcomes after noncardiac surgery: toward an empirical definition of hypotension. Anesthesiology. 2013 Sep;119(3):507-15. doi: 10.1097/ALN.0b013e3182a10e26. PMID 23835589
- [Background] Sudfeld S, Brechnitz S, Wagner JY, Reese PC, Pinnschmidt HO, Reuter DA, Saugel B. Post-induction hypotension and early intraoperative hypotension associated with general anaesthesia. Br J Anaesth. 2017 Jul 1;119(1):57-64. doi: 10.1093/bja/aex127. PMID 28974066
- [Background] Blokland Y, Farquhar J, Lerou J, Mourisse J, Scheffer GJ, Geffen GJ, Spyrou L, Bruhn J. Decoding motor responses from the EEG during altered states of consciousness induced by propofol. J Neural Eng. 2016 Apr;13(2):026014. doi: 10.1088/1741-2560/13/2/026014. Epub 2016 Feb 9. PMID 26859192
- [Background] Aho AJ, Kamata K, Jantti V, Kulkas A, Hagihira S, Huhtala H, Yli-Hankala A. Comparison of Bispectral Index and Entropy values with electroencephalogram during surgical anaesthesia with sevoflurane. Br J Anaesth. 2015 Aug;115(2):258-66. doi: 10.1093/bja/aev206. Epub 2015 Jul 1. PMID 26137969
- [Background] Sepulveda P, Cortinez LI, Irani M, Egana JI, Contreras V, Sanchez Corzo A, Acosta I, Sitaram R. Differential frontal alpha oscillations and mechanisms underlying loss of consciousness: a comparison between slow and fast propofol infusion rates. Anaesthesia. 2020 Feb;75(2):196-201. doi: 10.1111/anae.14885. Epub 2019 Dec 1. PMID 31788791
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Fudickar A, Kluzik A, Weiler N, Scholz J, Tonner PH, Bein B. A comparison of auditory evoked potentials derived from a monitor integrated module versus standard technique. J Neurosurg Anesthesiol. 2009 Apr;21(2):120-6. doi: 10.1097/ANA.0b013e3181990d00. PMID 19295390
- [Background] Ferreira AL, Mendes JG, Nunes CS, Amorim P. [Evaluation of Bispectral Index time delay in response to anesthesia induction: an observational study]. Braz J Anesthesiol. 2019 Jul-Aug;69(4):377-382. doi: 10.1016/j.bjan.2019.03.008. Epub 2019 Jul 29. PMID 31371175
- [Background] Zhong Q, Chen X, Zhao Y, Liu R, Yao S. Association of Polymorphisms in Pharmacogenetic Candidate Genes with Propofol Susceptibility. Sci Rep. 2017 Jun 13;7(1):3343. doi: 10.1038/s41598-017-03229-3. PMID 28611364
- [Background] Fan J, Zhou Q, Li Y, Song X, Hu J, Qin Z, Tang J, Tao T. Profiling of Long Non-coding RNAs and mRNAs by RNA-Sequencing in the Hippocampi of Adult Mice Following Propofol Sedation. Front Mol Neurosci. 2018 Mar 23;11:91. doi: 10.3389/fnmol.2018.00091. eCollection 2018. PMID 29628875
- [Background] Hallqvist L, Martensson J, Granath F, Sahlen A, Bell M. Intraoperative hypotension is associated with myocardial damage in noncardiac surgery: An observational study. Eur J Anaesthesiol. 2016 Jun;33(6):450-6. doi: 10.1097/EJA.0000000000000429. PMID 26950081